CLINICAL TRIAL: NCT02635672
Title: An Open-label, Multicenter Phase I Dose Escalation Study to Characterize Safety, Tolerability, Preliminary Anti-tumor Activity, Pharmacokinetics and Maximum Tolerated Dose of VIP152 (BAY 1251152) as Monotherapy or Combination Therapy in Subjects With Advanced Cancer.
Brief Title: Phase I Dose Escalation Study for VIP152 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vincerx Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VNC-152-101; 2014-004808-30 (EudraCT Number)
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Neoplasms
Keywords: Solid tumors; Aggressive non-hodgkin's lymphoma (NHL); Advanced Ovarian Cancer; Triple Negative Breast Cancer; DHL; Double-Hit Lymphoma; Transformed Follicular Lymphoma; Mantle Cell; Prostate Cancer; Melanoma; Non-small Cell Lung Cancer; Head and Neck Squamous Cell Cancer; Esophageal Cancer; Urothelial Carcinoma; Tumor Mutational Burden-High Cancer; Cutaneous Squamous Cell Carcinoma; Microsatellite Instability-High or Mismatch Repair Deficient Cancer; Microsatellite Instability-High or Mismatch Repair Deficient Colorectal Cancer; Gastric Cancer; Cervical Cancer; Hepatocellular Carcinoma; Merkel Cell Carcinoma; Renal Cell Carcinoma; Endometrial Carcinoma; MYC overexpression; MYC amplification; MYC translocation; Classic Hodgkins; Primary Mediastinal Large B Cell Lymphoma
MeSH Terms: conditions — Neoplasms; Triple Negative Breast Neoplasms; Prostatic Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Carcinoma, Transitional Cell; Stomach Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Merkel Cell; Carcinoma, Renal Cell; Endometrial Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose escalation of VIP152 (BAY 1251152) / PART 1 (Completed) (Experimental): Investigating VIP152 (BAY 1251152) in a dose escalation cohort in patients with solid tumors and aggressive NHL
  Interventions: Drug: VIP152 (BAY 1251152)
- Dose expansion of VIP152 (BAY 1251152) / PART 2 (Experimental): Investigating VIP152 (BAY 1251152) in a dose expansion cohort in patients with solid tumors and aggressive NHL
  Interventions: Drug: VIP152 (BAY 1251152) 30 mg
- Dose escalation of VIP152 (BAY 1251152) in combination with Keytruda® (pembrolizumab) / PART 3 (Experimental): Investigating combination VIP152 (BAY 1251152) and Keytruda® (pembrolizumab) in a dose escalation cohort in patients with advanced cancer. All subjects must be eligible to use pembrolizumab per USPI.
  Interventions: Drug: Keytruda; Drug: VIP152 (BAY 1251152) 15 mg
- Dose expansion of VIP152 (BAY 1251152) in combination with Keytruda® (pembrolizumab) / PART 4 (Experimental): Investigating combination VIP152 (BAY 1251152) and Keytruda® (pembrolizumab) in a dose expansion cohort in patients with advanced cancer. All subjects must be eligible to use pembrolizumab per USPI.
  Interventions: Drug: VIP152 (BAY 1251152) 30 mg; Drug: Keytruda

INTERVENTIONS:
Drug: VIP152 (BAY 1251152) — The starting dose of Cohort 1 will be 5 mg IV (30 minute infusion) fixed dose once weekly (5 mg/week) for 21 day cycles.
  Arms: Dose escalation of VIP152 (BAY 1251152) / PART 1 (Completed)
Drug: VIP152 (BAY 1251152) 30 mg — 30 mg IV (30 minute infusion) fixed dose once weekly of a 21 day cycle.
  Arms: Dose expansion of VIP152 (BAY 1251152) / PART 2; Dose expansion of VIP152 (BAY 1251152) in combination with Keytruda® (pembrolizumab) / PART 4
Drug: Keytruda — 200 mg IV fixed dose once every 3 weeks of a 21 day cycle
  Other Names: pembrolizumab
  Arms: Dose escalation of VIP152 (BAY 1251152) in combination with Keytruda® (pembrolizumab) / PART 3; Dose expansion of VIP152 (BAY 1251152) in combination with Keytruda® (pembrolizumab) / PART 4
Drug: VIP152 (BAY 1251152) 15 mg — The starting dose of Cohort 3 will be 15 mg IV (30 minute infusion) fixed dose once weekly (15 mg/week) for 21 day cycles.
  Arms: Dose escalation of VIP152 (BAY 1251152) in combination with Keytruda® (pembrolizumab) / PART 3

SUMMARY:
Determine the safety, tolerability, pharmacokinetics, maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of VIP152 (BAY 1251152) as monotherapy or in combination in patients with solid tumors and aggressive non-hodgkin's lymphoma (NHL).

DETAILED DESCRIPTION:
Part 2 VIP152 Monotherapy (Global). Part 3 dose escalation with VIP152 in combination with pembrolizumab (US only). Part 4 dose expansion with VIP152 in combination with pembrolizumab (US only).

ELIGIBILITY:
Part 2 (Global), Part 3 (US Only), and Part 4 (US Only)

Inclusion Criteria:

* Male or female patients aged >/=18 years
* Patients with a histologically or cytologically confirmed solid tumor or aggressive NHL who are refractory to or have exhausted all available therapies with MYC expression or known C-MYC amplification/alterations
* Adequate bone marrow, liver, and renal functions
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2

In the addition to the above Part 3 (US Only) and Part 4 (US Only)

* Must be eligible to use pembrolizumab per USPI

Exclusion Criteria:

* Active clinically serious infections of events > Grade 2
* Subjects who have new or progressive brain or meningeal or spinal metastases.
* Anticancer chemotherapy or immunotherapy during the study or within 1 weeks prior to the first dose of study drug
* Major surgery or significant trauma within 4 weeks before the first dose of study drug
* Allogeneic bone marrow transplant or stem cell rescue within 4 months before first dose of study drug; patients must have completed immunosuppressive therapy before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-02-10 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Incidence of DLT (Dose limit toxicity) of VIP152 (BAY1251152) | Cycle 1 Day 1 through Cycle 2 Day 1, where each cycle is up to 21 days
Maximum observed drug concentration in measured matrix after single dose administration (Cmax) of VIP152 (BAY1251152) | Cycle 1 Day 1 through Cycle 2 Day 1, where each cycle is up to 21 days
Area under the concentration versus time curve from zero to infinity after single (first) dose (AUC) of VIP152 (BAY1251152) | Cycle 1 Day 1 through Cycle 2 Day 1, where each cycle is up to 21 days
AUC from time 0 to the last data point > Lower limit of quantitation (LLOQ) [AUC(0-tlast)] of VIP152 (BAY1251152) | Cycle 1 Day 1 through Cycle 2 Day 1, where each cycle is up to 21 days
Maximum observed drug concentration in measured matrix after multiple dose administration during a dosage interval (Cmax,md) of VIP152 (BAY1251152) | Cycle 1 Day 1 through Cycle 2 Day 1, where each cycle is up to 21 days
AUC from time 0 to the last data point > LLOQ after multiple dosing [AUC(0-tlast)md] of VIP152 (BAY1251152) | Cycle 1 Day 1 through Cycle 2 Day 1, where each cycle is up to 21 days
Recommended phase 2 dose (RP2D) of VIP152 (BAY 1251152) | Cycle 1 Day 1 through Cycle 2 Day 1, where each cycle is up to 21 days
Incidence of DLT (Dose limit toxicity) of VIP152 (BAY1251152) in combination with Keytruda® (pembrolizumab) | Cycle 1 Day 1 through Cycle 3 Day 1, where each cycle is up to 21 days
Recommended phase 2 dose (RP2D) of VIP152 (BAY 1251152) in combination with Keytruda® (pembrolizumab) | Cycle 1 Day 1 through Cycle 2 Day 1, where each cycle is up to 21 days
Number of participants with adverse events as a measure safety and tolarability | Cycle 1 Day 1 up to 30 days after the last dose, where each cycle is up to 21 days (up to approximately 36 months)

SECONDARY OUTCOMES:
Tumor response evaluation based on the response criteria as applicable (RECIST v1.1 criteria for solid tumors and revised Lugano Classification for aggressive NHL) | Up to 3 Cycle 1 Day 1 up to 30 days after the last dose, where each cycle is up to 21 days (up to approximately 36 months)

CONTACTS AND LOCATIONS:
Overall Officials: Vincerx Study Director, Study Director — Vincerx Pharma, Inc.
Locations (16):
- United States (13):
  - Highlands Oncology Group, Springdale, Arkansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Maryland Oncology Hematology, Silver Spring, Maryland
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Willamette Valley Cancer Institute, Eugene, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Avera Health, Sioux Falls, South Dakota
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - NEXT Oncology, Austin, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
- Chile (2):
  - Centro de Investigaciones Clínicas Viña del Mar, Viña del Mar, Región de Valparaíso
  - Oncocentro, Viña del Mar
- START Madrid- Fundación Jiménez Diaz, Madrid, Spain

REFERENCES:
- [Derived] Diamond JR, Boni V, Lim E, Nowakowski G, Cordoba R, Morillo D, Valencia R, Genvresse I, Merz C, Boix O, Frigault MM, Greer JM, Hamdy AM, Huang X, Izumi R, Wong H, Moreno V. First-in-Human Dose-Escalation Study of Cyclin-Dependent Kinase 9 Inhibitor VIP152 in Patients with Advanced Malignancies Shows Early Signs of Clinical Efficacy. Clin Cancer Res. 2022 Apr 1;28(7):1285-1293. doi: 10.1158/1078-0432.CCR-21-3617. PMID 35046056
- See also: Click here and search for information on any recalls, market or product safety alerts by the FDA which might have occurred with this product. — https://www.fda.gov/drugs/drug-safety-and-availability